CLINICAL TRIAL: NCT00184106
Title: A Randomised, Triple Blind, Placebo-controlled Trial Comparing the Effects of Cognitive Therapy, Paroxetine and Both Cognitive Therapy and Paroxetine in the Treatment of Patients With Primary Social Phobia
Brief Title: RCT of Cognitive Therapy, Paroxetine, Combined CT and Paroxetine and Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: SP/NTNU-2005
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Phobic Disorders
Keywords: Phobic disorders; Therapy, cognitive; Paroxetine
MeSH Terms: conditions — Phobic Disorders | interventions — Paroxetine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Therapy (Active Comparator): Cognitive Therapy
  Interventions: Drug: Seroxat, Cognitive therapy, Seroxat+ cognitive therapy
- Seroxat and SE (Active Comparator): SSRI with Self exposure
  Interventions: Drug: Seroxat, Cognitive therapy, Seroxat+ cognitive therapy
- Seroxat and Cognitive Therapy (Active Comparator): Combination of Seroxat and Cognitive Therapy
  Interventions: Drug: Seroxat, Cognitive therapy, Seroxat+ cognitive therapy
- Pill-Placebo (Placebo Comparator): Pill Placebo
  Interventions: Drug: Seroxat, Cognitive therapy, Seroxat+ cognitive therapy

INTERVENTIONS:
Drug: Seroxat, Cognitive therapy, Seroxat+ cognitive therapy — Seroxat was administered over 24 weeks 20-50 mg/d, and Cognitive therapy was provided over 12 weeks. The patients were assessed at pre, post and 1 yrs follow up
  Other Names: Paroxetine

SUMMARY:
We aim to (1) evaluate the effectiveness of cognitive therapy and paroxetine and their combination, (2) investigate the patterns of change and the mechanisms of action involved during treatment by using psycho-physiological assessments in order to delineate some of the cognitive, behavioural and physiological mechanisms in the patients' response to CT, to paroxetine and placebo.One hundred patients with a primary diagnosis of social phobia will be selected and randomised into four treatment conditions. The first group (N=25) will be treated with CT alone, the second group (N=25) with CT plus paroxetine, the third group (N=25) with paroxetine and clinical management (TAU), the fourth group will receive placebo and clinical management (N=25). All patients will have 12 weeks of treatment in the acute phase, which includes 12 sessions of individual treatment for the two first groups. The 2nd and 3rd groups will in addition have 12 weeks of drug treatment in the maintenance phase. The 4th group will have placebo for 24 weeks and clinical management. The patients will be assessed at pre-treatment, at 12 weeks and at the end of treatment of the acute phase (12 weeks) and by the end of maintenance phase (24 weeks). Follow-up will be at 6 and 12 months.

Measures are based on all three main sources; self-report inventories, clinical assessments by independent raters and psycho-physiological assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to entry in the study.
2. Diagnosed with primary social phobia, generalized or specific (DSM-IV, APA, 1994).
3. Symptoms present at least one year.
4. Age between 18-65 years.

Exclusion Criteria:

1. Known somatic diseases.
2. Pregnant (*) or lactating women.
3. Psychosis
4. Acute suicidal symptoms
5. Major depressive disorder
6. Generalized Anxiety Disorder or PTSD
7. Cluster A or cluster B personality disorder
8. Substance abuse or dependence
9. Body dysmorphic disorder.
10. Not willing to accept random allocation.
11. Patients who take some form of SSRI medications currently or during the last 6 months
12. Patients not willing to withdraw psychotropic medication for a period of 4 weeks prior to entry to the trial or are taking herbal remedies that may be hazardous or inflict treatment response.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The proportion responders as measured by FAIR OF NEGATIVE EVALUATION and SPAI at 12 and 24 week. | December 2010
A patient is classified as responder if the decrease on FNE is equivalent with or above 40%. | December 2010

SECONDARY OUTCOMES:
Relapse rate during 6 and 12 months of follow up. | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Hans M Nordahl, Professor, Principal Investigator — Norwegian University of Science and Technology, NTNU
Locations (1):
- Dept. of Psychology, NTNU, Trondheim, Dragvoll, Norway

REFERENCES:
- [Result] Nordahl HM, Vogel PA, Morken G, Stiles TC, Sandvik P, Wells A. Paroxetine, Cognitive Therapy or Their Combination in the Treatment of Social Anxiety Disorder with and without Avoidant Personality Disorder: A Randomized Clinical Trial. Psychother Psychosom. 2016;85(6):346-356. doi: 10.1159/000447013. Epub 2016 Oct 15. PMID 27744447
- [Result] Nordahl H, Nordahl HM, Hjemdal O, Wells A. Cognitive and metacognitive predictors of symptom improvement following treatment for social anxiety disorder: A secondary analysis from a randomized controlled trial. Clin Psychol Psychother. 2017 Nov;24(6):1221-1227. doi: 10.1002/cpp.2083. Epub 2017 Mar 15. PMID 28295802